CLINICAL TRIAL: NCT03068559
Title: Consequences of an Initial Treatment for Head and Neck Cancer on Swallowing Function: Impact on Nutritional Status
Acronym: DYSPHAGIA
Status: Completed | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/05; 2012-A01030-43 (Other: ANSM ID RCB)
Record Dates: First submitted 2017-02-15; First posted 2017-03-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2017-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: * Patient must have an initial confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx.
  * Patient has to be aged ≥ 18
  * Patient has to be able to complete questionnaire in French
  * Patient must benefit from health insurance
  * Patient must sign an informed consent form
  * Patient treatment must be validated in a medical multidisciplinary team meeting: surgery, radiotherapy (RT), chemotherapy (CT), radiochemotherapy (RTCT), induction chemotherapy followed by radiochemotherapy (IND+RTCT), surgery followed by radiotherapy (surgery+RT), surgery followed by radiochemotherapy (surgery+RTCT).

SUMMARY:
The aim of the present prospective study was to assess dysphagia (occurrence, severity, length) in head and neck cancer (HNC), from diagnosis to 18 months after their first line treatment regardless of the treatment. The investigators have complied with the pre-listed clusters.

For this purpose, pursuant to consensus on the dysphagia assessment, the investigators used the Deglutition Handicap Index (DHI) questionnaire (Silbergleit 2012) for dysphagia screening and patient's self-perception. This was the only questionnaire validated in French evaluating the swallowing function by the patient (Woizard 2006).

Clinical evaluation according to NCI-CTCAE v4.0 criteria and objective measures of swallowing function were also recorded and compared to DHI results.

DETAILED DESCRIPTION:
Swallowing is one of the main functions in which oral, pharyngeal and laryngeal functions cooperate. Tumors in this area, as well as their treatments, can seriously impair the swallowing function, inducing dysphagia, a common complication still badly diagnosed. However, its impact is constant and always negative on the nutritional status, the treatment feasibility and the patients' quality of life.

Many teams have tried to determine assessment tools, prevalence and dysphagia treatment strategies. Thus, recently, in 2014, Kraaijenga et al. made a systematic review of the literature on these topics. Only 19 studies had been selected on the two previous years. Out of them, 7 were also literature reviews, including Raber-Durlacher's paper listing all dysphagia publications from 1990 to 2010. In the other 12 selected studies, 9 were prospective ones but with either a small number of patients or a specific treatment focused (e.g. Intensity Modulation Radiation Therapy, radiochemotherapy). For the dysphagia assessment, Kraaijenga et al. concluded that there is a need for simple self-evaluation scales compared to professional evaluation ones. The recording of some global indicators of functional status such as weight, dietary changes, nutritional tube dependence, is also advised. They concluded that patient-reported measures were commonly applied and provided complementary perspectives.

More recently, in 2015, Schlinder et al. reported a consensus proposition on the management of swallowing difficulties in head and neck patients treated by radiotherapy, that was discussed in the 2013 Milan congress. Six clusters of statements about these difficulties were reached related to: 1 and 2/ the assessment scales: one patient-reported -the MD Anderson Dysphagia Inventory- and one operator-reported outcome scales -NCI CTCAE criteria; 3/ the risk factors: research of signs and symptoms of dysphagia consequences e.g. aspiration; 4/ a preventive swallowing dysfunction evaluation (nutritionist and deglutologist evaluation); 5/ radiotherapic precautions; 6/ Preventive and therapeutic swallowing exercises.

The aim of the present prospective study was to assess dysphagia (occurrence, severity, length) in head and neck cancer (HNC), from diagnosis to 18 months after their first line treatment regardless of the treatment. The investigators have complied with the pre-listed clusters.

For this purpose, pursuant to consensus on the dysphagia assessment, the investigators used the Deglutition Handicap Index (DHI) questionnaire (Silbergleit 2012) for dysphagia screening and patient's self-perception. This was the only questionnaire validated in French evaluating the swallowing function by the patient.

Clinical evaluation according to NCI-CTCAE v4.0 criteria and objective measures of swallowing function were also recorded and compared to DHI results.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have an initial confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx.
* Patient has to be aged ≥ 18
* Patient has to be able to complete questionnaire in French
* Patient must benefit from health insurance
* Patient must sign an informed consent form
* Patient treatment must be validated in a medical multidisciplinary team meeting: surgery, radiotherapy (RT), chemotherapy (CT), radiochemotherapy (RTCT), induction chemotherapy followed by radiochemotherapy (IND+RTCT), surgery followed by radiotherapy (surgery+RT), surgery followed by radiochemotherapy (surgery+RTCT).

Exclusion Criteria:

* - Patients treated with prior systemic chemotherapy, radiation therapy or surgery on head and neck area
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a HNCC beginning a first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
moderate to severe dysphagia | 18 months
  DHI questionnaire

SECONDARY OUTCOMES:
frequency of dysphagia reported by investigator using NCI-CTCAE v4.0 grading | 18 months
comparison of grade 2 to 4 clinical dysphagia and self-perceived moderate/severe dysphagia | 18 months
  (DHI questionnaire, score ≥16)
time of dysphagia occurrence | 18 months
length of dysphagia | 18 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 18 months
necessity and total length of Enteral Nutrition | 18 months

IPD SHARING:
Plan to Share IPD: No